CLINICAL TRIAL: NCT05532293
Title: A Phase I, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose and Multiple Ascending Dose Clinical Study to Assess the Safety, Tolerability and Pharmacokinetics of MSP008-22 in Healthy Adult Volunteers
Brief Title: Phase One Clinical Trial to Assess the Safety, Tolerability and Pharmacokinetics of MSP008-22 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Godavari Biorefineries Limited (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Clinexel-GBL-003; CTRI/2022/08/045056 (Other: Clinical Trials Registry-India)
Record Dates: First submitted 2022-09-05; First posted 2022-09-08 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: COVID-19
Keywords: Single Ascending Dose; Phase 1; Multiple Ascending Dose; randomised, double blind; MSP008-22; healthy volunteers; COVID-19; safety; tolerability; pharmacokinetics
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Phase I, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose and Multiple Ascending Dose Clinical Study to Assess the Safety, Tolerability and Pharmacokinetics of the Investigational Product in Healthy Adult Volunteers
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Both the Investigator and study participants will remain blinded to the treatment administered (drug or placebo) till the final results of the study are obtained.
  The placebo will identical to the investigational medicinal product in smell, taste, and appearance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSP008-22 (Experimental): MSP008-22 is a New Chemical Entity (NCE) that has demonstrated positive outcomes during in vitro and in vivo studies for COVID19.
  Formulated as tablets intended for oral dosing to trial participants.
  Interventions: Drug: MSP008-22
- Placebo (Placebo Comparator): placebo will be identical in smell, taste, and appearance to the tablets of MSP008-22
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MSP008-22 — MSP008-22 is a small molecule with demonstrated anticancer activity in-vitro & in vivo studies. As several anticancer drugs are also good antiviral drugs, it was anticipated that MSP008-22 can also be a promising anti-COVID drug. Accordingly, in vitro assay studies and in an in vivo study in golden Syrian hamster were conducted where MSP008-22 has shown good anti-SARSCoV2 effects.MSP008-22.
  Arms: MSP008-22
Other: Placebo — Placebo tablets identical in appearance, taste and smell to the tablets of MSP008-22
  Arms: Placebo

SUMMARY:
This is a Phase I clinical study of MSP008-22, the Investigational Medicinal Product (IMP). The current study is designed to evaluate the safety and tolerability and pharmacokinetics of single and multiple oral doses of the IMP (MSP008-22) in healthy volunteers.

DETAILED DESCRIPTION:
MSP008-22 is a New Chemical Entity (NCE) that has demonstrated positive outcomes during in vitro and in vivo studies for COVID19.

This clinical study is planned as a double blind, randomised, placebo-controlled, combined clinical study of two parts: Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) studies, respectively. Pharmacokinetic (PK) profile of the MSP008-22 will also be assessed in both parts of the study. The safety, tolerability and pharmacokinetic data and results obtained from this study will determine the potentially efficacious doses of the IMP (MSP008-22) in the subsequent efficacy studies in COVID-19 patients.

The SAD Part will consist of 6 cohorts of 8 healthy adult volunteers, each volunteer will be randomly (blinded) allocated to MSP008-22 or placebo (each cohort will consist of 6 volunteers receiving MSP008-22 and 2 volunteers receiving placebo). Six (6) dose levels (200 (OD), 400(OD), 400(BD), 600(BD), 800(BD) and 1000 (BD) mg) of MSP008-22 are selected for oral administration. An additional cohort of 8 volunteers (6:2 MSP008-22 vs placebo) of lower doses of MSP008-22 (less than 1000 mg BD) may be recruited into the SAD Part, if required.

The MAD Part will consist of 2 cohorts of 8 healthy adult volunteers, each volunteer will be randomly (blinded) allocated to MSP008-22 or placebo (each cohort will consist of 6 volunteers receiving MSP008-22 and 2 volunteers receiving placebo). Two (2) dose levels (800(BD) and 1000(BD) mg) of the MSP008-22 are selected for oral administration.

An additional cohort of 8 volunteers (6:2 MSP008-22 vs placebo) of lower doses of MSP008-22 (less than 1000 mg BD) may be recruited into the MAD Part, if required.

Healthy adult volunteers eligible for participations in the study will be enrolled as study participants. They will be randomly assigned to the study drug (MSP008-22) and placebo arm during both the SAD and MAD parts of the study.

A total of eighty (80) healthy adult volunteers volunteer (48 in the 06 cohorts of SAD part and 16 in the 02 cohorts of MAD part, and 16 subjects of the 02 additional cohorts in either SAD or MAD part of the study, if required) are planned to be enrolled and randomized in the study.

Between each cohort, an interim analysis of PK, safety and tolerability will be performed. An independent Drug Safety Monitoring Board (DSMB) will provide recommendations about stopping, modifying or continuing the study. Decision to escalate to next higher dose level/ Ccohort will be based on interim analysis of pharmacokinetic data, safety data at 36-hr post-dose, as well as during the safety follow-up of 30-days post dose. Once a particular dose level is judged to be safe by the DSMB, the study will proceed and doses administered to the study subjects will escalate to the next higher dose level/ cohort.

The dosing and the conduct of study between the cohorts will be staggered by approximately 2 to 4 weeks.

Both the Investigator and study participants will remain blinded to the treatment administered (drug or placebo) till the final results of the study are obtained.

Safety evaluation during both the SAD & MAD pars of the clinical study will include adverse events, clinical laboratory/ pathological test results, electrocardiogram (ECG), and measurement of vital signs.

Blood samples for pharmacokinetic profiling of MSP008-22 will be collected as follows:

* for the first 04 dose cohorts of the SAD Part of the Study - at pre-dose (30 min prior to dosing), and at 1h, 2h, 4h, 8h, 12h, and 24h, and 36 h.
* for the last 02 dose cohorts of the SAD Part of the Study - at pre-dose (30 min prior to dosing), and at 1h, 1.5h, 2h, 3h, 4h, 8h, 12h (pre dose for 2nd dose (approx. 02 mins prior to 2nd dose)), 14h, 16h, 18h, 24.00, and 36h.
* for Day 1 of MAD part of the Study - at pre-dose (30 min prior to dosing), 1h, 1.5h, 2h, 3h, 4h, 8h, 12h (pre dose for 2ndpre dose (approx. 02 mins prior to 2nd dose)), 14h, 16h, 18h, and 24h (pre dose for 1st dose for Day 2 (approx. 02 mins prior to Day-2-1st dose)).
* For Day 2 of MAD part of the Study - sample collected at 24h after Day 1-1st dose will be serve the purpose of pre-dose sample for Day 2 1st dose).
* For Days 3 - 6 of MAD part of the Study - at pre-dose (30 mins prior to dosing of 1st dose/ morning dose).
* for Day 7 of MAD part of the Study - at pre-dose (30 min prior to dosing), 1h, 1.5h, 2h, 3h, 4h, 8h, 12h (pre dose for 2nd dose (approx. 02 mins prior to 2nd dose)), 14h, 16h, 18h, 24h and 36h.

ELIGIBILITY:
Inclusion Criteria:

Volunteers will be enrolled in the study when the following inclusion criteria will be met:

1. Should be healthy adult volunteer in the age range of 18-50 years old (both inclusive).
2. Should be healthy adult volunteers, with a BMI 18-30 kg/m2 (both inclusive).
3. Volunteer is able to read the volunteer information sheet, to understand information about the study and willing to sign the informed consent voluntarily.
4. Healthy as determined by pre-study medical history, physical examination, vital signs, haematology, chemistry parameters, pulse rate and/or blood pressure, and ECG within the reference range, or showing no clinically relevant deviations, as judged by the Investigator.
5. Negative tests for Hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (anti-HCV) and human immunodeficiency virus (HIV)-l and HIV -2 antibody at screening.
6. Clinical laboratory test results clinically acceptable at screening and admission.
7. Negative screen for alcohol and drugs of abuse at screening and admission.
8. Non-smokers or ex-smokers (must have ceased smoking >12 months prior screening visit). If a former smoker, reason for stopping smoking to be investigated.
9. The volunteer must agree to comply with the drawing of blood samples for the PK assessments.
10. The volunteer is willing and able to comply with all testing and requirements defined in the protocol.
11. The volunteer is willing and able to remain at the study site for the duration of the confinement period as per the protocol requirements or if exceeded, on Investigator's discretion, if exceeded and return for the outpatient visit.

    If female:
12. Woman with no childbearing potential by reason of surgery or at least 1-year post-menopause (Le., 12 months post last menstrual period), or menopause confirmed by follicle-stimulating hormone (FSH) testing;
13. If of childbearing potential, using an effective nonhormonal method of contraception· (intrauterine device or intrauterine system; condom or occlusive cap [diaphragm or cervical or vault caps] with spermicidal foam or gel or film or cream or suppository; true abstinence; or vasectomized male partner, provided that he is the sole partner of that volunteer) for all the duration of the study and up to one month after the last Investigational medicinal product (IMP) administration;
14. Negative serum pregnancy test at screening and negative urine pregnancy test on admission of each treatment period (women of childbearing potential only);

    If Male
15. Using an effective method of contraception (condom or occlusive cap [diaphragm or cervical or vault caps] with spermicidal foam or gel or film or cream or suppository; true abstinence; or vasectomy) throughout the study and up to one month after the last IMP administration

Exclusion Criteria:

Volunteers meeting any of the following criteria will be excluded from this clinical study:

1. The volunteer has any relevant deviations from normal in physical examination, electrocardiogram (ECG), or clinical laboratory tests, as evaluated by the Investigator.
2. The volunteer has had a clinically significant illness or conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs, within 30 days of Check-in for the study.
3. The volunteer has a clinically relevant history or presence of significant respiratory, neurological, hepatic, renal, endocrine, cardiovascular, neurological, gastrointestinal, pulmonary, haematological, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue, lymphatic or metabolic disease or disorders.
4. The volunteer has a significant infection or known inflammatory process on screening or admission.
5. The volunteer has acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhoea, heartburn) at the time of screening or admission.
6. The volunteer has a clinically significant surgical history
7. The volunteer has used any prescription medication within 14 days of dosing or over-the-counter (OTC) medication within 48 h of dosing or intends to use any prescription medication or OTC medication during the study that may interfere with the evaluation of study medication.
8. The volunteer has had used medicines within 2 weeks of admission that may affect the safety or other study assessments, in the investigator's opinion
9. The volunteer has consumed alcohol, caffeine or xanthine-containing products 48 h before dosing or intends to use any of these products during the study.
10. The volunteer has consumed grapefruit, grapefruit juice, or grapefruit-containing products 7 days before dosing or intends to use any of these products during the study.
11. The volunteer has a history of substance abuse or a positive ethanol breath test, urine cotinine, or urine drug screen at screening or at check-in.
12. The volunteer has a positive HIV test at the Screening Visit.
13. The volunteer has received an investigational drug within 30 days of Check-in.
14. Use of any investigational drug within 30 days, or 5 half-lives, whichever is longer, prior to the planned first drug administration.
15. The volunteer has participated in more than 2 clinical studies within the 12 months prior to screening.
16. The volunteer has used any investigational drug or participated in any clinical trial within 90 days prior to dosing in this study.
17. The volunteer has donated or lost a significant volume of blood (>450 mL) within 4 weeks prior to the study.
18. The volunteers have a history of hyperemesis
19. The volunteer is unwilling to reside in the study site for the duration of the study or to cooperate fully with the investigator or site personnel.
20. The volunteer has an AST/ALT or total bilirubin greater than the ULN. One repeat test will be allowed.
21. The volunteer has a history of relevant atopy or drug hypersensitivity or known intolerance to the inactive ingredients in the IMP.
22. The volunteer has clinically relevant abnormalities found in physical examination, vital signs measurements, laboratory safety tests or ECG, e.g. QTc according to Bazett: QTc > 450ms, PQ > 220ms, QRS > 120ms
23. The volunteer has supine pulse rate not within 45 to 90 beats per minute and/or supine blood pressure Systolic < 90 >145 mmHg and diastolic < 40 > 95 mmHg.
24. Surgery or trauma with significant blood loss within 2 months before the planned screening for the trial.
25. Any social and medical condition that would jeopardize the volunteer's appropriate participation in this study.
26. Have any medical dietary restrictions.
27. Cannot communicate reliably with the Investigator(s)
28. Are unlikely to co-operate with the requirements of the study.
29. Known or suspected of not being able to comply with the trial protocol and/or clinical unit restrictions.
30. Are unwilling or unable to give written informed consent.
31. Volunteer is an employee of the Sponsor, the Investigator or the Institution of the Investigator.

    If female:
32. Pregnancy or breast-feeding.
33. Woman of childbearing potential not using an accepted effective contraceptive method or using oral contraceptives

    If male:
34. Not using an accepted effective method of contraception.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events [Time Frame- ] | 30 days post last dose for each cohort
  To assess safety & tolerability of MSP008-22 in Human
Incidence of serious adverse events (SAEs) by relation to the IMP (related/not related) | 30 days post last dose for each cohort
  To assess safety & tolerability of MSP008-22 in Human
Percentage of volunteers who experience at least 1 Treatment Emergent Adverse Event (TEAE) | 30 days post last dose for each cohort
  To assess safety & tolerability of MSP008-22 in Human
Percentage of volunteers who discontinue due to an Adverse Event (AE). | 30 days post last dose for each cohort
  To assess safety & tolerability of MSP008-22 in Human
Percentage of volunteers who meet the markedly abnormal criteria for safety laboratory tests at least once post dose. | 7 days post last dose for each cohort
  To assess safety MSP008-22 in Human
Percentage of volunteers who meet the markedly abnormal criteria for vital sign measurements at least once post dose | 7 days post last dose for each cohort
  To assess safety MSP008-22 in Human
Percentage of volunteers who meet the markedly abnormal criteria for safety electrocardiogram (ECG) parameters at least once post dose. | 7 days post last dose for each cohort
  To assess safety MSP008-22 in Human

SECONDARY OUTCOMES:
Plasma Cmax | post-dose in Single ascending Dose trial & post dose on days 1 & 7 in Multiple ascending dose part of the trial
  Maximum plasma concentrations
Plasma Tmax | post-dose in Single ascending Dose trial & post dose on days 1 & 7 in Multiple ascending dose part of the trial
  Time to Maximum plasma concentrations (tmax)
Plasma AUC0-t | Single ascending Dose
  Area under the concentration-time curve from dosing (time 0) to time t [AUC0-t]
Plasma AUC0-inf | Single ascending Dose
  Area under the concentration-time curve from dosing (time 0) extrapolated to infinite time [AUC 0-inf]
Plasma AUC0-tau | post dose on days 1 & 7 in Multiple ascending dose part of the trial
  Area under the concentration-time curve to the end of the dosing period [AUC 0-tau]
Plasma AUC0-t | post dose on day 7 in Multiple ascending dose part of the trial
  Area under the concentration-time curve from dosing (time 0) to time t [AUC0-t]
Plasma Kel | in Single ascending Dose trial & post-dose on day 7 in Multiple ascending dose part of the trial
  Elimination constant [Kel]
Plasma t1/2 | in Single ascending Dose trial & post dose on day 7 in Multiple ascending dose part of the trial
  Elimination half life [t1/2]
Plasma Ctrough | on days 2 & 6 in Multiple ascending dose part of the trial
  Pre-dose plasma trough concentration (Ctrough)
Plasma Racc | post dose on days 1 & 7 in Multiple ascending dose part of the trial
  Accumulation ratio Racc (Cmax on Day 7/Cmax on Day 1), (AUC0-τ on Day 7/AUC0-τ on Day 1) and (Ctrough on Day 7/Ctrough on Day 1)

CONTACTS AND LOCATIONS:
Overall Officials: Deepa Arora, MD, Study Director — Clinexel Life Sciences Pvt. Limited
Locations (2):
- India (2):
  - K. J. Somaiya Hospital & Research Centre, Somaiya Ayurvihar Complex, Eastern Express Highway, Sion East, Mumbai, Maharashtra
  - Ashirwad Hospital & Research Centre, Maratha Section, Near Jijamata Udyan, Ulhasnagar, Maharashtra, India, Ulhasnagar, Maharashtra

IPD SHARING:
Plan to Share IPD: No